CLINICAL TRIAL: NCT06315179
Title: Seattle Spatial Transcriptomic Research in Inflammatory Bowel Disease Evaluation
Brief Title: Seattle Spatial Transcriptomic Research in Inflammatory Bowel Disease Evaluation (STRIDE)
Acronym: STRIDE
Status: Recruiting | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Allen Institute (Unknown)
Responsible Party: Principal Investigator, Betty Zheng, Assistant Professor, Director of Advanced IBD Fellowship Program, Seattle Children's Hospital
Other Study IDs: STUDY00004616
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Indeterminate Colitis; Functional Abdominal Pain Syndrome; Functional Bowel Disorder; Esophageal Diseases; Gastroduodenal Disorder; Bowel Dysfunction; Gallbladder Diseases; Sphincter of Oddi Dysfunction; Anorectal Disorder
Keywords: IBD; DGBI
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Esophageal Diseases; Intestinal Diseases; Gallbladder Diseases; Sphincter of Oddi Dysfunction; Rectal Diseases | interventions — Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — -The blood and tissue bio-specimens obtained for this research will undergo genetic testing including but not limited to single-cell analysis, exome sequencing, and whole genome sequencing, gene editing, and organoid generation (results will not be provided to participants and/or their care providers). Cells are not 'immortalized' and will eventually expire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Inflammatory Bowel Disease: Participants will enroll before their initial diagnostic procedure. After pathology results are reported, participants will be categorized based on the assigned diagnoses: Inflammatory Bowel Disease (IBD) [Crohn's disease (CD), ulcerative colitis (UC), and Indeterminate Colitis (IC)] vs Disorders of the Brain-Gut Interactions (DGBI).
  Participation in the IBD cohort will last for three years.
  Interventions: Diagnostic Test: Esophagogastroduodenoscopy (EGD) with biopsy; Diagnostic Test: Colonoscopy w/ biopsy
- Disorders of the Brain-Gut Interactions: Participants will enroll before their initial diagnostic procedure. After pathology results are reported, participants will be categorized based on the assigned diagnoses: Inflammatory Bowel Disease (IBD) [Crohn's disease (CD), ulcerative colitis (UC), and Indeterminate Colitis (IC)] vs Disorders of the Brain-Gut Interactions (DGBI).
  -The DGBI cohort will be subdivided into: Esophageal Disorder, Gastroduodenal Disorder, Bowel Disorder, Centrally Mediated Disorders of GI Pain, Gallbladder and Sphincter of Oddi Disorder, Anorectal Disorder, Childhood Functional GI Disorders: Neonate/Toddler, Childhood Functional GI Disorders: Child/Adolescent
  Participation in the DGBI cohort will include the initial sample and data collection as well an one further medical record extraction at month 24.
  Interventions: Diagnostic Test: Esophagogastroduodenoscopy (EGD) with biopsy; Diagnostic Test: Colonoscopy w/ biopsy

INTERVENTIONS:
Diagnostic Test: Esophagogastroduodenoscopy (EGD) with biopsy — Esophagogastroduodenoscopy (EGD) is a test procedure to examine the lining of the esophagus, stomach, and first part of the small intestine.
Diagnostic Test: Colonoscopy w/ biopsy — Colonoscopy is a test procedure to examine the lining of the different portions of the large intestine: cecum, colon, rectum, and anal canal.

SUMMARY:
This is a prospective observational study collecting long-term clinical data and samples for research in pediatric inflammatory bowel disease (IBD) patients with gut inflammation and a control cohort of pediatric patients with disorders of the brain-gut interactions (DBGI) with no detectable gut inflammation.

DETAILED DESCRIPTION:
Research procedures will coincide with clinical visits at institutional standards. As part of their clinical disease evaluation, participants will have blood, stool, and tissue collected as indicated by their disease course. Additional research samples or data will be collected during these visits. Participants will be asked to collect urine samples specifically for research.

ELIGIBILITY:
Inclusion Criteria:

* Suspected diagnosis of CD (Crohn's Disease), UC (Ulcerative Colitis) or Indeterminate colitis (IC)

Exclusion Criteria:

* Evidence of Other Complicating Medical Issues:
* Other serious medical conditions, such as neurological, liver, kidney, or systemic disease
* Pregnancy
* Tobacco, alcohol, or illicit drug abuse

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All individuals who meet inclusion criteria will be approached.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Bio-repository sample collection for spatial transcriptomics | 3 years
  Collection of blood and stool samples at baseline month 1, month 2, month 3, month 6, month 12, month 24, and month 36. Tissue will be collected at baseline and at any follow-up endoscopy or surgical intervention.

SECONDARY OUTCOMES:
Paris Classification of Crohn's Disease | Baseline
  * Age at diagnosis
  * Location of disease: distal 1/3 +- ileum limited cecal disease, colonic, ileocolonic, upper disease proximal to ligament of treitz, upper disease distal to ligament of treitz and proximal to distal 1/3 ileum
  * Behavior of disease: non-stricturing/non-penetrating, stricturing, penetrating, both penetrating and stricturing disease, either at the same or different times
  * Perianal sub type: yes, no, do not know
  * Growth sub type: no evidence of growth delay, growth delay
Montreal Classification of Crohn's disease | Baseline
  * Age at diagnosis
  * Location of disease: terminal ileal +- limited cecal disease, colonic, ileocolonic, isolated upper disease
  * Behavior of disease: non-stricturing/non-penetrating, stricturing, penetrating, both penetrating and stricturing disease, either at the same or different times
Paris Classification of Ulcerative Colitis/Indeterminate Colitis | Baseline
  * Extent of disease: ulcerative proctitis, left-sided UC (distal to splenic flexure), extensive (hepatic flexure distally), pancolitis (proximal to hepatic flexure)
  * Severity: never severe, ever severe
Montreal Classification of Ulcerative Colitis/Indeterminate Colitis | Baseline
  * Extent of disease: ulcerative proctitis, left-sided UC (distal to splenic flexure), extensive (proximal to splenic flexure)
  * Severity: clinical remission, mild UC, moderate UC, severe UC
Disorder of Gut-Brain Interaction classification | Baseline
  Diagnoses super-type and applicable sub type:
  * Esophageal Disorders
  * Gastroduodenal Disorder
  * Bowel Disorder
  * Centrally Mediated Disorders of GI Pain
  * Gallbladder and Sphincter of Oddi Disorder
  * Anorectal Disorder
  * Childhood Functional GI Disorders: Neonate/Toddler
  * Childhood Functional GI Disorders: Child/Adolescent
Physician's Global Assessment (PGA) | 3 years
  Severity: Quiescent, Mild, Moderate, Severe

CONTACTS AND LOCATIONS:
Overall Officials: Betty (Hengqi) Zheng, MD, Principal Investigator — Seattle Children's Hospital, University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No